CLINICAL TRIAL: NCT04998084
Title: Understanding the Importance of the Microbiome and Metabolome in IBD Patients
Brief Title: Advanced Therapy Registry of IBD Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Eli Sprecher, MD, Director of Clinical Research and Development Department, Tel-Aviv Sourasky Medical Center
Other Study IDs: 0162-19-TLV
Record Dates: First submitted 2021-06-27; First posted 2021-08-10 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Crohn Disease; Ulcerative Colitis; Pouchitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Pouchitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is aim to detect common microbial profiles and metabolic pathways throughout IBD diagnosis and treatment with biological therapy.

DETAILED DESCRIPTION:
The study is aim to detect common microbial profiles and metabolic pathways in patients belonging to the following groups:

1. Therapy naïve newly diagnosed Crohn's disease (CD), ulcerative colitis (UC) and pouchitis patients. Studying this group of patients will enable the detection of microbial profiles associated with disease onset.
2. Patients planned to commence biological therapy (with or without IBD). Studying this group of patients will enable the detection of microbial profiles associated with response to biological therapy.
3. IBD patients in complete remission (treated or untreated with biologics). Following this group of patients will enable the detection of microbial profiles associated with disease exacerbation.

Methods:

Study design: A prospective cohort study. Setting: The investigators will prospectively collect clinical, behavioral and environmental data of patients participating in the study. Data will be collected according to a uniform standardized protocol specifically adapted to the needs of the study and shared between the collaborators.

Study population: Eligible patients, who sign an informed consent form and answer to all the study inclusion criteria. Patients will be informed of the study by their treating physician, recruited and followed throughout the follow-up period by study coordinators.

sample size: sample size was estimated according to clinical capabilities of the researcher. We aim to collect data from a total of 1000 patients.

Schedule: Data will be collected between the years 2019-2024.

Study plan:

Patient and disease characteristics At baseline, demographic characteristics, medical history and specifically IBD phenotype, severity, extent and location, disease duration, previous medicinal treatment will be documented. Baseline and follow-up study visits which will include biological sample collection and questionnaires.

Patients will be asked to complete questionnaires to account for their lifestyle, sleep, quality of life and disease related symptoms and outcomes. Physician global assessment (PGA), disease severity using clinical scores (HBI and SCCAI scores for CD and UC patients) and biochemical data (CRP, fecal calprotectin) will be documented.

ELIGIBILITY:
Inclusion Criteria:

Patients who belong to one of the following sub-groups:

1. Newly diagnosed (<1 years), therapy naïve IBD and pouchitis patients
2. IBD patients in complete remission (treated or untreated with biologics)
3. Patients (with and without IBD) scheduled to commence a biological therapy

Exclusion Criteria:

1. Age≤18 years
2. Inability to sign an informed consent
3. Abdominal surgery during the previous 3 months
4. Systemic antibiotic therapy in the previous 4 weeks
5. Severe systemic disease such as kidney, liver, neurologic, cardio-vascular disease
6. Primary sclerosing cholangitis
7. Pregnancy at recruitment
8. Cancer within the previous 5 years excluding local NMSC

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigators aim to collect data from a total of 1000 patients.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2024-06-27 (Estimated); Study Completion 2025-06-27 (Estimated)

PRIMARY OUTCOMES:
Clinical response as determined by a decrease in Harvey-Bradshaw Index (HBI) or Simple Clinical Colitis Activity Index (SCCAI) decrease of ≥3 points among CD and UC patients respectively. | 2019-2024
Biologic response as determined by a decrease in C-Reactive Protein (CRP), fecal calprotectin >10% from baseline. | 2019-2024
Improvement in patient quality of sleep score | 2019-2024
  as determined by a decrease of >10% from baseline.
Improvement in patient quality of life score | 2019-2024
  as determined by a decrease of >10% from baseline.
Improvement in stress score | 2019-2024
Clinical response as determined by the Harvie Bradshaw Index (HBI)>3 points among crohn's patients | 2019-2024
Clinical response as determined by the Simple Clinical Colitis Activity Index (SCCAI)>3 points among UC patients | 2019-2024

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided